CLINICAL TRIAL: NCT07024186
Title: Soft Tissue Augmentation by Xenogenic Collagen Matrix Versus Sub Epithelial Connective Tissue Graft Around Early Implant Placement in Maxillary Esthetic Zone
Brief Title: Xenogenic Collagen Matrix vs. Connective Tissue Graft for Soft Tissue Augmentation Around Early Maxillary Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Omar ismail phd, PhD Candidate, Faculty of Dentistry, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Study ID: 505-2021
Record Dates: First submitted 2025-05-12; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Alveolar Bone Loss; Gingival Recession; Peri-implant Mucositis
Keywords: Xenogenic Collagen Matrix; Connective Tissue Graft; Soft Tissue Augmentation
MeSH Terms: conditions — Alveolar Bone Loss; Gingival Recession

STUDY DESIGN:
Intervention Model Description: Participants are assigned in parallel to either the xenogeneic collagen matrix group or the subepithelial connective tissue graft group for soft tissue augmentation around early implant placement in the maxillary esthetic zone. Group allocation is determined by simple randomization using a coin toss.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor responsible for evaluating soft tissue volume and esthetic results is blinded to the group allocation to reduce assessment bias. Participants and care providers are not blinded due to the nature of the surgical interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xenogeneic Collagen Matrix (Active Comparator): This arm involves the use of a xenogeneic collagen matrix for soft tissue augmentation around early implant placement in the maxillary esthetic zone.
  Interventions: Procedure: Xenogeneic Collagen Matrix
- Subepithelial Connective Tissue Graft (Active Comparator): This arm involves the use of a subepithelial connective tissue graft for soft tissue augmentation around early implant placement in the maxillary esthetic zone.
  Interventions: Procedure: subepithelial connective tissue graft

INTERVENTIONS:
Procedure: Xenogeneic Collagen Matrix — Xenogeneic Collagen Matrix The xenogeneic collagen matrix is a biomaterial used to promote soft tissue regeneration and support healing in dental implant procedures.
  Arms: Xenogeneic Collagen Matrix
Procedure: subepithelial connective tissue graft — ubepithelial Connective Tissue Graft The subepithelial connective tissue graft is a biological tissue taken from the patient's own palate or other donor sites to promote healing and aesthetic outcomes around dental implants.
  Arms: Subepithelial Connective Tissue Graft

SUMMARY:
This study compares two methods used to improve gingival tissue around dental implants placed in (the maxillary esthetic zone). After a tooth is removed and a dental implant is placed early (usually 4-8 weeks later), additional soft tissue is sometimes needed to ensure the implant looks natural and functions well. The two techniques being studied are:

Subepithelial connective tissue graft (SCTG) - where tissue is taken from the patient's own mouth (usually the palate)

Xenogeneic collagen matrix (XCM) - a processed collagen material from animals, used as a substitute for the patient's own tissue.

The goal is to see which method is better in terms of gingival thickness, esthetic appearance, healing, and patient comfort. This research may help dentists choose the most effective and comfortable treatment for their patients.

DETAILED DESCRIPTION:
Dental implants in the anterior maxillary region (esthetic zone) are commonly used to replace missing teeth. When implants are placed using the early placement protocol (typically 4-8 weeks after tooth extraction), additional soft tissue volume may be required to ensure an esthetically pleasing and functionally stable result.

Soft tissue augmentation can be achieved using:

Subepithelial connective tissue grafts (SCTG): A technique that involves harvesting tissue from the patient's own palate and placing it around the implant to improve gingival thickness and contour.

Xenogeneic collagen matrix (XCM): A biocompatible, animal-derived collagen scaffold designed to substitute for autologous tissue, reducing patient morbidity and surgical time.

This study is a prospective, randomized, controlled, parallel-arm clinical trial conducted at Minia University, Faculty of Dentistry. Eligible patients missing a single tooth in the anterior maxilla with a thin gingival biotype and requiring early implant placement were recruited. A total of 20 patients were randomly assigned into two groups (10 per group):

Group 1 (Control): Received subepithelial connective tissue graft harvested from the palate using the single-incision technique.

Group 2 (Test): Received xenogeneic collagen matrix (Mucoderm®) adapted and inserted into the grafting site.

Outcome Measures:

Primary Outcome:

Change in gingival thickness (GT) at 12 months post-surgery, measured via transgingival probing using a standardized protocol.

Secondary Outcomes:

Change in width of keratinized tissue (KTW)

Esthetic outcome (using clinical photographs and standardized scoring systems, e.g., Pink Esthetic Score)

Post-operative healing and complications

Patient-reported outcomes regarding comfort, pain, and satisfaction (using Visual Analog Scale questionnaires)

Clinical and radiographic assessments were performed at baseline, 6 months, and 12 months post-implant placement.

Ethical approval was obtained from the Research Ethics Committee of Minia University, and all participants provided informed consent. The study adheres to the Declaration of Helsinki and ICH-GCP guidelines.

This research aims to provide evidence on whether xenogeneic collagen matrix can serve as a viable, less invasive alternative to autogenous tissue grafts in implant dentistry, especially for cases with esthetic demand and thin soft tissue biotype.

ELIGIBILITY:
**Inclusion Criteria:**

* Non-restorable or hopeless teeth from maxillary anterior to first premolar due to one or more of the following:
* Extensive caries
* Root fractures
* Inability to perform functional crown lengthening due to gingival zenith line with high gingival display
* Improper crown-to-root ratio due to bone removal leading to aesthetic or restorative failure
* Patients aged 25-55 years
* Both male and female patients
* Thin tissue biotype

**Exclusion Criteria:**

* Pregnant women
* Smokers
* Presence of persistent chronic infection at the implant site
* Patients in the growth phase with partially erupted teeth
* Patients with parafunctional habits such as bruxism or clenching that may overload the implant
* Patients with insufficient vertical inter-arch space in centric occlusion to accommodate restorative components

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Peri-implant soft tissue thickness | 12 months after implant placement
  change in soft tissue thickness measured in millimeters at the buccal aspect of the implant site.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed O Ismail, MSc, Principal Investigator — Faculty of Dentistry, Minia University
Locations (1):
- Minya, Minya, Minya Governorate, Egypt

DOCUMENTS (2):
  • Study Protocol (2021-07-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT07024186/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT07024186/SAP_001.pdf